CLINICAL TRIAL: NCT05326282
Title: A Proof of Concept Study Evaluating the Role of Emerging Ultrasound Technologies in the Assessment and Monitoring of Localised Prostate Cancer in Men on an Active Surveillance Programme
Brief Title: Evaluating the Role of Ultrasound in Prostate Cancer
Acronym: ERUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: R2706
Record Dates: First submitted 2021-09-06; First posted 2022-04-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer
Keywords: Ultrasound; Micro-ultrasound; Active surveillance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Men with suspected or low grade prostate cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-parametric and micro ultrasound (Experimental): Transrectal ultrasound imaging in men with suspected or known low grade prostate cancer using both standard and micro-ultrasound technology
  Interventions: Diagnostic Test: Multi-parametric ultrasound

INTERVENTIONS:
Diagnostic Test: Multi-parametric ultrasound — Diagnostic ultrasound parameters used to evaluate the prostate. Transrectal scans will be performed
  Other Names: Micro-ultrasound

SUMMARY:
Active surveillance (AS) is becoming an increasingly common treatment option for men who have been diagnosed with localised low-grade prostate cancer (PCa). Low-grade disease is commonly noted by clinicians to be clinically insignificant cancer but remains a psychological burden to many men in this cohort. There is consensus that regular review is required for men on AS so that early treatment can be undertaken if there is disease progression, and to support men living with a cancer diagnosis. Some AS protocols, including National Institute for Clinical Excellence (NICE), advocate the use of MRI as a regular part of the monitoring pathway.

Unfortunately, access to MRI for AS, within the current health care environment in the UK, is limited due to increasing demand for primary diagnostic examinations, particularly in the post pandemic recovery phase. Emerging technologies in ultrasound imaging may, however, add another diagnostic tool to monitor disease for patients on AS. This proof of concept study is to evaluate whether new multi-parametric ultrasound techniques can safely reduce the number of MRIs required for effective AS.

Men being investigated for PCa will be invited to undergo an ultrasound examination of their prostate, via the rectum, in addition to the diagnostic MRI undertaken as part of normal care. The findings of the ultrasound will be directly compared with the MRI and any subsequent biopsy samples taken as part of routine care. Those who then progress onto AS will be invited to undergo regular rectal prostate ultrasound examinations. These will be compared with previous imaging for signs of change.

This study will also evaluate the changing role of practitioners who will be using new technologies and making decisions about disease progression. The ability to implement new techniques will be assessed. All imaging will be undertaken at Castle Hill Hospital over a 24-month period from commencement of the study.

DETAILED DESCRIPTION:
Research Plan 1.1 Purpose and design Across the UK prostate cancer is the most common cancer in men. Developments in magnetic resonance imaging (MRI), and the implementation of a targeted biopsy regime, have resulted in a considerable improvement in the detection of prostate cancer.

1.1.1 Clinical context: Prostate cancer can be present as an indolent low-grade cellular change to the tissue but with very little risk of this progressing to a metastatic life threatening disease. Despite the improved diagnostic capabilities, there remain a significant proportion of men in whom low-grade cancer is detected and consequent treatment options may present a higher risk to quality of life than the presence of the localised disease. Both active surveillance (AS) and watchful waiting (WW) involve proactively monitoring the patient for signs of disease progression rather than undertaking treatment immediately.

The improvements in MRI imaging and reporting indicate that regular scans would add valuable information for patients under AS but capacity is significantly hindering this as an available application.

1.1.2 Technological improvements Emerging technologies in ultrasound imaging, which is less hindered by capacity issues within the UK and is utilised, to a degree, in current standard care, may add another diagnostic tool to monitor disease for patients on AS. A multi-parametric ultrasound assessment may provide the crucial diagnostic features that enables ultrasound imaging to be used to monitor disease. A crucial question remains as to whether the use of additional imaging and health care intervention could improve patient outcomes.

1.1.3 Normalisation Process Theory (NPT) Despite the publication of a defined framework for the development and evaluation of research, there remain substantial problems in the design and conduct of studies introducing complex interventions and their subsequent implementation. If a new technology provides good diagnostic results but is cumbersome and complex to use, it is unlikely to be implemented into routine healthcare practice. A recognised gap exists between developing new treatments and knowledge, and implementing these in practice for the patient who may benefit. An understanding of the ability to implement the proposed new complex ultrasound techniques in real-life clinical practice will be explored within this proof of concept study.

1.2 Study Aim This aim of this proof of concept study is to evaluate if emerging ultrasound technologies can provide reliable and reproducible imaging that can be used to assess the prostate gland in men with known localised prostate cancer and who are being managed with active surveillance.

As with many research studies, data is collected in a strict and controlled environment which may not readily translate into a real life clinical setting. The feasibility for implementing changes to the imaging pathways in active surveillance will also be evaluated with the clinical team delivering the current and future service.

1.3 Primary and secondary objectives 1.3.1 Primary objective The primary objective of the study is to evaluate if emerging multi-parametric ultrasound technologies can provide a viable tool to be used in the active surveillance of men with known localised prostate cancer.

1.3.2 Secondary objectives

Secondary objectives of this study are:

* to evaluate the diagnostic parameters of diagnostic ultrasound that can be utilised to assess disease within the prostate gland.
* To evaluate the diagnostic parameters of diagnostic ultrasound that can be utilised to assess disease progression within the prostate gland.
* To evaluate if the intra and inter operator variability in the assessment of ultrasound imaging parameters of the prostate gland can be investigated.
* To determine if a suitable standardise imaging protocol and reporting tool or model could be utilised in the reporting of transrectal ultrasound imaging of the prostate.
* To gain a better understanding of how new ultrasound technology and techniques can be implemented and embedded into clinical practice.

1.4 Study phases

This study is being undertaken as a doctorate research project but within the National Health Service (NHS) care setting. The study will consist of four phases:

1.4.1 Phase 1: In this initial phase, eligible men who have consented to participate will undergo a transrectal ultrasound examination with a standard ultrasound probe and, at the same attendance a transrectal ultrasound examination with a new and novel probe using 29MHz scanning frequency. The images obtained from this examination will be retrospectively compared with the MRI imaging that has been obtained as part of the standard care pathway. The images obtained will be reviewed by two health care practitioners with experience in prostate imaging and the outcomes of these reviews compared to evaluate agreement levels.

1.4.2 Phase 2: The second phase of the study will evaluate the use of multiparametric standard and micro ultrasound in the assessment of men who are on an AS or WW pathway. This phase the study will evaluate if there are any changes in the findings at repeat ultrasound examinations that can indicate disease progression. Eligible men, who have consented to participate, will again undergo a transrectal ultrasound examination with a standard ultrasound probe and, at the same attendance a transrectal ultrasound examination with a new and novel probe using 29 megahertz (MHz) scanning frequency.

1.4.3 Phase 3: The process and acceptability of implementing new interventions and technologies into everyday clinical practice is frequently overlooked following research trials. This third phase will explore the views of the health care practitioners, who have consented to participate, regarding the use and implementation of the proposed new technologies; skill mix between these professional groups will be required for successful long term practice. The participants will be recruited from differing professionals within the staff groups of Hull University Teaching Hospitals NHS Trust. An adapted survey tool, derived from normalisation process theory framework, will be used to better understand how and if the new, complex, multi-parametric ultrasound techniques can be implementation within the organisational setting of everyday routine practice. A baseline assessment of confidence in knowledge and skills related to prostate cancer evaluation using ultrasound will be made.

1.4.3.1 Staff training: Participants in phase 3 will then be provided with training using specific multi-parametric ultrasound (US) techniques and will regularly score multi-parametric US examinations. Participants' confidence in knowledge and skills, related to prostate cancer evaluation using US, and how the participants feel this technology can be implemented into regular patient care will be assessed, using the same adapted survey at baseline at 6 - 12 months' post implementation.

1.4.4 Phase 4: A fourth phase of the study is planned. Once outcomes from the initial 3 phases of the study are known the lead researcher intends to organise a national meeting where results will be presented and discussion held between the research team and other centres providing a diagnostic prostate cancer service. The aim of this event is to disseminate results and to obtain a wider understanding of its acceptance beyond local practice. Multi-parametric ultrasound is novel and there may be resistance to wider implementation. Opportunities and barriers will be explored at this phase 4 event.

ELIGIBILITY:
Inclusion Criteria:

* he recruitment criteria and pathway for the clinical phases of the study are outlined in the flow charts, appendix 1 and appendix 2. These identify when the participants will be invited to participate, when consent will be obtained and the broad outline of the involvement in the study that participants can expect.

Inclusion criteria for phase 1

Men referred to urology within Hull University Teaching Hospitals NHS Trust with suspected, but undiagnosed, prostate cancer and:

* Age equal to 75 or less
* PSA equal to 20 or less
* Life expectancy of 10 years or more
* Multi-parametric MRI performed as part of routine care pathway
* Are able to tolerate a rectal ultrasound examination
* Able to provide informed consent to the study

Inclusion criteria for phase 2

Men referred to urology within Hull University Teaching Hospitals NHS Trust with known localised prostate cancer of Gleason 3 + 3 (6) or less and:

* Are eligible for an AS monitoring pathway
* Are on an AS monitoring pathway which is regularly reviewed by a consultant urologist
* Able to attend Castle Hill Hospital for 6 monthly multi-parametric US examinations
* Are able to tolerate a rectal ultrasound examination
* Able to provide informed consent to the study

Inclusion criteria for phase 3

* Health care practitioner working as a radiologist or sonographer and employed within radiology of Hull University Teaching Hospitals NHS Trust
* Hold a recognised qualification awarded by the Royal College of Radiologists or a recognised post graduate ultrasound qualification undertaken at a consortium for accreditation of sonographic education (CASE) approved higher education institute
* Registered with a statutory regulator such as the General Medical Council (GMC), Nursing and Midwifery Council (NMC), Health and Care Professions Council (HCPC)
* Participates in the current radiology prostate cancer assessment care pathway
* Able to provide informed consent to the study

Exclusion Criteria:

* the recruitment criteria and pathway for the clinical phases of the study are outlined in the flow charts, appendix 1 and appendix 2. These identify when the participants will be invited to participate, when consent will be obtained and the broad outline of the involvement in the study that participants can expect.

Inclusion criteria for phase 1

Men referred to urology within Hull University Teaching Hospitals NHS Trust with suspected, but undiagnosed, prostate cancer and:

* Age equal to 75 or less
* PSA equal to 20 or less
* Life expectancy of 10 years or more
* Multi-parametric MRI performed as part of routine care pathway
* Are able to tolerate a rectal ultrasound examination
* Able to provide informed consent to the study

Inclusion criteria for phase 2

Men referred to urology within Hull University Teaching Hospitals NHS Trust with known localised prostate cancer of Gleason 3 + 3 (6) or less and:

* Are eligible for an AS monitoring pathway
* Are on an AS monitoring pathway which is regularly reviewed by a consultant urologist
* Able to attend Castle Hill Hospital for 6 monthly multi-parametric US examinations
* Are able to tolerate a rectal ultrasound examination
* Able to provide informed consent to the study

Inclusion criteria for phase 3

* Health care practitioner working as a radiologist or sonographer and employed within radiology of Hull University Teaching Hospitals NHS Trust
* Hold a recognised qualification awarded by the Royal College of Radiologists or a recognised post graduate ultrasound qualification undertaken at a CASE approved higher education institute
* Registered with a statutory regulator such as the GMC, NMC or HCPC
* Participates in the current radiology prostate cancer assessment care pathway
* Able to provide informed consent to the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male only as this study is specifically looking at the prostate gland which is absent in females
Enrollment: 100 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
The number of identified changes on ultrasound, within the prostate glands of participants, that correlate with changes identified on the gold standard active surveillance imaging | 24-Months from commencement of the study
  Ultrasound will be used to image the prostate in patients with suspected and known low grade prostate cancer. The ultrasound images will be compared with the gold standard of prostate MRI, and the histology, from any biopsy undertaken. The ultrasound images will be evaluated to assess for any changes to the appearance of the prostate to understand if prostate disease progression can be detected.

SECONDARY OUTCOMES:
Change in confidence and knowledge in users of new ultrasound techniques will be measured using a normalization process theory survey completed at baseline and at 12 months following implementation of the study. | 12-months from commencement of this study
  Staff using new technology and novel diagnostic parameters may be challenged by this different technique. Implementation into clinical practice may be difficult. This phase of the study will evaluate the barriers and opportunities the new technology can bring to staff working in this field

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Parker, MSc, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Ultrasound, Radiology, Hull, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised data will be shared. This will take the form of ultrasound images that have been stored with all identifiable data removed. The ultrasound images will be shared and available for review with other researchers

REFERENCES:
- [Background] Parker PC, Harrison G. Educating the future sonographic workforce: membership survey report from the British Medical Ultrasound Society. Ultrasound. 2015 Nov;23(4):231-41. doi: 10.1177/1742271X15605344. Epub 2015 Sep 29. PMID 27433263
- [Result] da Silva V, Cagiannos I, Lavallee LT, Mallick R, Witiuk K, Cnossen S, Eastham JA, Fergusson DA, Morash C, Breau RH. An assessment of Prostate Cancer Research International: Active Surveillance (PRIAS) criteria for active surveillance of clinically low-risk prostate cancer patients. Can Urol Assoc J. 2017 Aug;11(8):238-243. doi: 10.5489/cuaj.4093. PMID 28798822
- [Result] de Brun T, O'Reilly-de Brun M, O'Donnell CA, MacFarlane A. Learning from doing: the case for combining normalisation process theory and participatory learning and action research methodology for primary healthcare implementation research. BMC Health Serv Res. 2016 Aug 3;16(a):346. doi: 10.1186/s12913-016-1587-z. PMID 27488361
- [Result] Field LJ, Snaith BA. Developing radiographer roles in the context of advanced and consultant practice. J Med Radiat Sci. 2013 Mar;60(1):11-5. doi: 10.1002/jmrs.2. Epub 2013 Feb 5. PMID 26229602
- [Result] Finch TL, Girling M, May CR, Mair FS, Murray E, Treweek S, McColl E, Steen IN, Cook C, Vernazza CR, Mackintosh N, Sharma S, Barbery G, Steele J, Rapley T. Improving the normalization of complex interventions: part 2 - validation of the NoMAD instrument for assessing implementation work based on normalization process theory (NPT). BMC Med Res Methodol. 2018 Nov 15;18(1):135. doi: 10.1186/s12874-018-0591-x. PMID 30442094
- [Result] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Result] Klotz L, Vesprini D, Sethukavalan P, Jethava V, Zhang L, Jain S, Yamamoto T, Mamedov A, Loblaw A. Long-term follow-up of a large active surveillance cohort of patients with prostate cancer. J Clin Oncol. 2015 Jan 20;33(3):272-7. doi: 10.1200/JCO.2014.55.1192. Epub 2014 Dec 15. PMID 25512465

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT05326282/Prot_000.pdf
  • Informed Consent Form (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT05326282/ICF_001.pdf